CLINICAL TRIAL: NCT00121680
Title: A Phase I/Ib, Multicenter, Open-Label, Dose Escalation Study of E7080 in Patients With Solid Tumors and in Combination With Temozolomide in Patients With Advanced and/or Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-102
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Melanoma
Keywords: cancer
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7080

INTERVENTIONS:
Drug: E7080 — Oral.

SUMMARY:
The purpose of this study is to study the safety of E7080 administered to patients with solid tumors or lymphomas.

Please note: this study is now recruiting patients with advanced and/or metastatic melanoma only.

In the current phase of this study, To determine the MTD and the pharmacokinetic profile of E7080 when given as continuous daily (qd) dosing in combination with temozolomide.

ELIGIBILITY:
Inclusion Criteria:

Patients with a histologically and/or cytologically confirmed solid tumor or lymphoma who are resistant/refractory to approved therapies or for whom no curative therapies are available All previous treatment (including surgery and radiotherapy) must have been completed at least four weeks prior to study entry and any acute toxicities must have resolved Aged 18 years. Because of the potential additional risk to children suggested by preclinical models of dysplasia in growing epiphyseal growth plates, enrollment will be limited to adult patients ECOG performance status score of 0 or 1 Written informed consent prior to any study specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice Willing and able to comply with the protocol guidelines for the duration of the study For patients in the Schedule 2 Expanded Melanoma Cohort only: histologically and/or cytologically confirmed advanced and/or metastatic melanoma who are resistant/refractory to approved therapies or for whom no curative therapies are available. In addition, patients must have melanoma lesions amenable to tissue biopsy and must agree to undergo biopsies of malignant and adjacent non-malignant tissue pretreatment and at the end of Cycle 1 of treatment For patients in the Melanoma Combination Cohort only: histologically and/or cytologically confirmed melanoma that is advanced and/or metastatic

Exclusion Criteria:

Untreated or unstable metastases to the central nervous system (CNS) tumors. Patients who have completed local therapy and have discontinued the use of steroids for this indication at least 4 weeks prior to commencing treatment and in whom stability has been proven by at least 2 CT or MRI scans obtained at least 4 weeks apart are permitted Any of the following laboratory parameters: hemoglobin < 9 g/dL (5.6 mmol/L); neutrophils <1.5 x 109/L; platelets <100 x 109/L; serum bilirubin >25 mol/L (1.5 mg/dL); liver function tests with values >3 x upper limit of normal (ULN); renal function with serum creatinine >1.5 ULN or creatinine clearance < 60 mL/min Positive history of HIV, active hepatitis B or active hepatitis C or severe/uncontrolled intercurrent illness or infection Patients with centrally located non-small cell lung cancers and squamous cell lung cancers Clinically significant cardiac impairment or unstable ischemic heart disease including a myocardial infarction within six months of study start Patients with marked Baseline prolongation of QT/QTc interval (QTc interval > 450 msec for males or > 470 msec for females) using the Fridericia method for QTc analysis Bleeding or thrombotic disorders, or using therapeutic dosages of anticoagulants, such as warfarin. Occasional use of NSAIDs and antiplatelet agents such as aspirin, clopidogrel, aggrenox and dipyridamole are not considered exclusionary if taken <7 days per 28 days. However, if the patient requires chronic use (>/=7 days out of 28 days) of full doses of aspirin or NSAIDs then the patient is excluded. Concomitant antiplatelet agents and NSAIDs should be used with caution Requirement for chronic use of full dose aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) Poorly controlled hypertension (defined as requiring changes in any hypertensive regimen within 1 week three months of study entry) or patients diagnosed with hypertension based on repeat blood pressure measurements of >160/90 mmHg at Screening >1+ proteinuria on urine dipstick testing or 30 mg/dL A history of gastrointestinal malabsorption or having undergone surgery requiring gastrointestinal anastomoses within four weeks of starting therapy or who have not recovered from major surgery within three weeks of starting therapy History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the Investigator, would impair study compliance Any treatment with investigational drugs within 30 days before the start of the study Previous treatment with E7080 Known intolerance to temozolomide (or any of the excipients) Women who are pregnant or breast-feeding; women of childbearing potential with a positive pregnancy test at Screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception (including two forms of contraception, one of which must be a barrier method) in the opinion of the Investigator (revised per Amendment 04). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential Fertile males with female partners who are not willing to use contraception or whose female partners are not using adequate contraceptive protection Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2005-07; Primary Completion 2011-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of E7080 for two different schedules incorporating dose interruptions. | Every two cycles.

SECONDARY OUTCOMES:
Identify the dose limiting toxicities (DLT); explore safety and tolerability; determine pharmacokinetic profile; explore anti-tumor efficacy. | Every two cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Inc., Study Director — Eisai Limited
Locations (2):
- United States (2):
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Kurzrock R, Atkins J, Wheler J, Fu S, Naing A, Busaidy N, Hong D, Sherman S. Tumor marker and measurement fluctuations may not reflect treatment efficacy in patients with medullary thyroid carcinoma on long-term RET inhibitor therapy. Ann Oncol. 2013 Sep;24(9):2256-61. doi: 10.1093/annonc/mdt177. Epub 2013 May 14. PMID 23676418